CLINICAL TRIAL: NCT02813291
Title: Effects of Motor Imagery Practice Combined With Transcranial Direct Current Stimulation in the Learning of a Complex Motor Sequence in Young and Elderly Subjects
Brief Title: MI Practice and tDCS With Aging
Acronym: MISt
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 69HCL15_0719
Record Dates: First submitted 2016-06-22; First posted 2016-06-24 (Estimated); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Aging; Motor Learning
Keywords: Motor imagery; transcranial direct current stimulation; motor learning; aging
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Stimulation group (Young Stim) (Experimental): Subjects of the Stimulation groups (Young Stim and Elderly Stim) will receive in parallel an anodal tDCS of the primary motor cortex.
  Interventions: Device: tDCS
- Stimulation group (Elderly Stim) (Experimental): Subjects of the Stimulation groups (Young Stim and Elderly Stim) will receive in parallel an anodal tDCS of the primary motor cortex.
  Interventions: Device: tDCS
- Sham group (Young Sham) (Sham Comparator): Subjects of the Sham groups (Young Sham and Elderly Sham) will receive in parallel a sham tDCS of the primary motor cortex.
  Interventions: Device: sham tDCS
- Sham group (Elderly Sham) (Sham Comparator): Subjects of the Sham groups (Young Sham and Elderly Sham) will receive in parallel a sham tDCS of the primary motor cortex.
  Interventions: Device: sham tDCS

INTERVENTIONS:
Device: tDCS — All subjects will mentally repeat a complex finger sequence with the left hand, for 13 min:
  - Subjects of the Stimulation groups (Young Stim and Elderly Stim) will receive in parallel an anodal tDCS of the primary motor cortex.
  Arms: Stimulation group (Elderly Stim); Stimulation group (Young Stim)
Device: sham tDCS — All subjects will mentally repeat a complex finger sequence with the left hand, for 13 min:
  - Subjects of the Sham groups (Young Sham and Elderly Sham) will receive in parallel a sham tDCS of the primary motor cortex.
  Arms: Sham group (Elderly Sham); Sham group (Young Sham)

SUMMARY:
The mental repetition of movements - or motor imagery (MI) practice - facilitates motor learning. It allows avoiding fatigue that occurs during physical practice; this method is thus particularly interesting for elderly people. Transcranial direct current stimulation (tDCS) is a noninvasive method of neurostimulation during which a low direct current is applied to the brain via electrodes placed on the scalp. This method has been successfully used to enhance motor learning in both young and elderly subjects.

The main aim of this study is to assess the impact of MI practice combined with tDCS on the learning of a complex finger sequence, in young and elderly subjects.

For that purpose, young and elderly healthy subjects will be randomly assigned to Stimulation and Sham groups. There will thus be a total of four groups: Young Stim, Young Sham, Elderly Stim, and Elderly Sham.

All subjects will participate to three training sessions spread over five days, and a retention test one week after the third training session.

During training they will mentally repeat a complex finger sequence with the left hand, for 13 min:

* Subjects of the Stimulation groups (Young Stim and Elderly Stim) will receive in parallel an anodal tDCS of the primary motor cortex.
* Subjects of the Sham groups (Young Sham and Elderly Sham) will receive in parallel a sham tDCS of the primary motor cortex.

Immediately before (pretest) and after (posttest) each training session, as well as during the retention test, subjects will repeat the sequence as many times of possible, for 1 min. During these tests (pretests, posttests and retention test) electroencephalographic activity will be recorded to assess the Mu rhythm power.

ELIGIBILITY:
Inclusion Criteria:

* Being aged between 20 and 35 years for the young subjects / between 65 and 80 years for the elderly subjects
* For elderly subjects: Mini Mental State Examination (MMSE) ≥ 24
* Being a male or a female
* Being right handed
* Taking an effective method of contraception for the women of childbearing age
* Having signed the consent form
* Being registered with a social security scheme

Exclusion Criteria:

* Presenting a neurologic, psychiatric or motor trouble
* Practicing or having practiced at least 5 hours by week an activity involving a high manual dexterity (e.g. piano)
* Showing any contraindication to tDCS:

  * History of epilepsy
  * head trauma with loss of consciousness
  * Implanted material (pacemaker, surgical clips, metal specks in the skull, etc.)
  * Past neurosurgical intervention
  * Open sore on the scalp
  * Consumption of more than three glasses of alcohol daily
  * Use of drugs
  * Pregnancy (positive pregnancy test)

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2017-04-26 (Actual); Primary Completion 2019-03-22 (Actual); Study Completion 2019-03-22 (Actual)

PRIMARY OUTCOMES:
Change in the number of correct sequences between first pretest and retention test | The number of correct sequences will be assessed at pretest of the first training session (day 1) and at retention test (day 10).
  Change will be calculated using the following formulae: (number of correct sequences at retention test - number of correct sequences at first pretest) / number of correct sequences at first pretest × 100

SECONDARY OUTCOMES:
Change in the number of correct sequences between first pretest and third posttest | The number of correct sequences will be assessed at pretest of the first training session (day 1) and at posttest of the third training session (day 3)
  Change will be calculated using the following formulae: (number of correct sequences at third posttest - number of correct sequences at first pretest) / number of correct sequences at first pretest × 100
Change in the power of the Mu rhythm between first pretest and retention test | The power of the Mu rhythm will be assessed at pretest of the first training session (day 1) and at retention test (day 10)
  Change will be calculated using the following formulae: (power of the Mu rhythm at retention test - power of the Mu rhythm at first pretest) / power of the Mu rhythm at first pretest × 100
Change in the power of the Mu rhythm between first pretest and third posttest | The power of the Mu rhythm will be assessed at pretest of the first training session (day 1) and at posttest of the third session (day 3)
  Change will be calculated using the following formulae: (power of the Mu rhythm at third posttest - power of the Mu rhythm at first pretest) / power of the Mu rhythm at first pretest × 100

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Krolak-Salmon, Pr, PU-PH, Principal Investigator — Hospices Civils de Lyon - Hôpital des Charpennes
Locations (1):
- Hospices Civils de Lyon - Hôpital des Charpennes - 27, rue Gabriel Péri, Villeurbanne, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Metais A., Muller C., Breuil C., Boublay N., di Rienzo F., Guillot A., Collet C., Krolak-Salmon P., Saimpont A. (2020). P143 Effects of Anodal tDCS combined with motor imagery on motor sequence learning in older adults. Clinical Neurophysiology 131(4):e93-e94. https://doi.org/10.1016/j.clinph.2019.12.254
- [Background] Muller C., Breuil C., Boublay N., Metais A., di Rienzo F., Guillot A., Collet C., Krolak-Salmon P., Saimpont A. (2020). P47 Effects of motor imagery and anodal tDCS on motor sequence learning in healthy young adults. Clinical Neurophysiology 131(4):e38-e39. https://doi.org/10.1016/j.clinph.2019.12.158